CLINICAL TRIAL: NCT00341965
Title: Pesticide Exposure and Health Status in NC African American Male Farmers and Farm Workers
Brief Title: Pesticide Exposure and Health Status in North Carolina African American Male Farmers and Farm Workers
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999006; OH99-E-N006
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2013-11-04

CONDITIONS: Pesticide Exposure
Keywords: DDT; DDE; Androgen Levels; Farming; Antiandrogen

SUMMARY:
We propose to conduct a study to increase our understanding of farming practices and of the potential for previous exposure to DDT in North Carolina African American male agricultural workers, a group especially likely to have had high DDT exposure. Because of potentially widespread DDT exposure from agricultural activities, African American farmers and farm workers may be uniquely at risk for any associated health effects. However, little is known about levels of pesticide exposure in African American farming populations. Three hundred and eighty-nine African American men who are current or former farmers or farm workers will be asked to participate in the study. These men are members of the Supplemental Minority Cohort of the NCI/NIEHS/EPA Agricultural Health Study (AHS). The AHS is a prospective study of the potential health effects associated with agricultural exposures. Men in the supplemental cohort were recruited in 1996. At that time, they completed an enrollment questionnaire that focused on lifetime agricultural exposures, demographics, lifestyle factors and health. In this new study, a follow-up questionnaire will be administered by telephone by a trained interviewer to all men. Following the interview, the participant will be asked to donate a blood specimen, to have anthropometric indices (e.g., height, weight, waist and hip circumference, etc.) measured, and to have a top- and side view Polaroid photograph of their head taken during one visit to a central community location, such as the local church or health clinic. We will quantitatively document serum p,p'-DDE levels, correlate these with self-reported farming activities and DDT exposure, and describe the health status of these men. We will also correlate serum p,p'-DDE levels and androgen concentrations, since p,p'-DDE is thought to be a potent androgen receptor antagonist. This exploration of the potential link between levels is important because the demonstration of any subclinical physiological effects of p,p'-DDE would increase the plausibility of a wide range of health effects that have been postulated to be associated with the endogenous endocrine environment and the so-called endocrine disrupters. In addition, we will evaluate the relationship between several important physiological parameters which can be easily and accurately measured in serum, and physical characteristics including hair patterning and distribution of body fat in these African American men.

DETAILED DESCRIPTION:
We propose to conduct a study to increase our understanding of farming practices and of the potential for previous exposure to DDT in North Carolina African American male agricultural workers, a group especially likely to have had high DDT exposure. Because of potentially widespread DDT exposure from agricultural activities, African American farmers and farm workers may be uniquely at risk for any associated health effects. However, little is known about levels of pesticide exposure in African American farming populations. Three hundred and eighty-nine African American men who are current or former farmers or farm workers will be asked to participate in the study. These men are members of the Supplemental Minority Cohort of the NCI/NIEHS/EPA Agricultural Health Study (AHS). The AHS is a prospective study of the potential health effects associated with agricultural exposures. Men in the supplemental cohort were recruited in 1996. At that time, they completed an enrollment questionnaire that focused on lifetime agricultural exposures, demographics, lifestyle factors and health. In this new study, a follow-up questionnaire will be administered by telephone by a trained interviewer to all men. Following the interview, the participant will be asked to donate a blood specimen, to have anthropometric indices (e.g., height, weight, waist and hip circumference, etc.) measured, and to have a top- and side view Polaroid photograph of their head taken during one visit to a central community location, such as the local church or health clinic. We will quantitatively document serum p,p'-DDE levels, correlate these with self-reported farming activities and DDT exposure, and describe the health status of these men. We will also correlate serum p,p'-DDE levels and androgen concentrations, since p,p'-DDE is thought to be a potent androgen receptor antagonist. This exploration of the potential link between levels is important because the demonstration of any subclinical physiological effects of p,p'-DDE would increase the plausibility of a wide range of health effects that have been postulated to be associated with the endogenous endocrine environment and the so-called endocrine disrupters. In addition, we will evaluate the relationship between several important physiological parameters which can be easily and accurately measured in serum, and physical characteristics including hair patterning and distribution of body fat in these African American men.

ELIGIBILITY:
* INCLUSION CRITERIA:

All African American men who are members of the Supplemental Minority Cohort of the NCI/NIEHS/EPA Agricultural Health Study will be recontacted and asked to participate in the study.

EXCLUSION CRITERIA:

We are limiting this initial study to adult African American males.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 1999-01-27; Study Completion 2013-11-04

CONTACTS AND LOCATIONS:
Overall Officials: Dale Sandler, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Alavanja MC, Sandler DP, McMaster SB, Zahm SH, McDonnell CJ, Lynch CF, Pennybacker M, Rothman N, Dosemeci M, Bond AE, Blair A. The Agricultural Health Study. Environ Health Perspect. 1996 Apr;104(4):362-9. doi: 10.1289/ehp.96104362. PMID 8732939
- [Background] Bagatell CJ, Bremner WJ. Androgens in men--uses and abuses. N Engl J Med. 1996 Mar 14;334(11):707-14. doi: 10.1056/NEJM199603143341107. No abstract available. PMID 8594431
- [Background] Austin SG, Huang N, Woernle CW. PMR study of mortality among Alabama workers and farmers. Am J Ind Med. 1995 Jan;27(1):29-36. doi: 10.1002/ajim.4700270104. PMID 7900733